CLINICAL TRIAL: NCT05558566
Title: Neurofeedback From the Supplementary Motor Area for Tourette Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000033043; 1R01MH127147-01A1 (NIH)
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Tourette Syndrome in Adolescence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback from the SMA (Experimental)
  Interventions: Other: Neurofeedback from the SMA
- Neurofeedback from control region (Active Comparator)
  Interventions: Other: Neurofeedback from control region

INTERVENTIONS:
Other: Neurofeedback from the SMA — Feedback is provided regarding activity in the SMA and participant attempts to control SMA activity using the feedback as a training signal
  Arms: Neurofeedback from the SMA
Other: Neurofeedback from control region — Feedback is provided regarding activity in a control region and participant attempts to control activity in that region using the feedback as a training signal.
  Arms: Neurofeedback from control region

SUMMARY:
This is a clinical trial where adolescents aged 10-16 years old with Tourette Syndrome (or chronic tic disorder) are randomized to receive either real-time functional magnetic resonance imaging (fMRI) neurofeedback targeting the supplementary motor area (for the experimental intervention) or real-time fMRI neurofeedback (NF) from a control region (for the control intervention).

DETAILED DESCRIPTION:
The training portion of this study involves three fMRI NF sessions, with six NF scans per session. NF scans alternate between up-regulate and down-regulate blocks in which participants are cued to increase or decrease activity in the target region while receiving feedback on activity in the region at the bottom of the screen in the form of a line graph. The experimental group receives feedback from the supplementary motor area (SMA) and the control group receives feedback from a control region of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls, 10 to 16 years of age
* A current diagnosis of Tourette Syndrome (TS) or chronic tic disorder (CTD), with active tics that can be executed without head movement, and a YGTSS score of at least 13 (for TS participants) or at least 12 (for CTD participants)
* Currently stable medication treatment and no planned changes in medication for the duration of the study.
* Family residence within 2 hours of Yale Medical Center with ability and willingness to attend assessment and fMRI visits.
* Children and their parents are expected to be able to speak and understand spoken English in order to participate in a clinical assessment of TS and related psychopathology.
* Subjects will be free of: 1) metal medical implants or braces, 2) pregnancy, and will have 3) a body weight of less than 250 lbs. and 4) no claustrophobia.

Exclusion Criteria:

* Intelligence quotient below 80
* Current diagnosis of autism spectrum disorder, bipolar or psychotic disorder or current suicidality
* Significant medical condition such as heart disease, hypertension, liver or renal failure, pulmonary disease, seizure disorder
* Recently initiated psychotherapy. Participation in the study will not be allowed within 8 weeks of the initiation of psychotherapy. Ongoing, concurrent psychotherapy (that was initiated at least 8 weeks previously) for the child will be allowed, but parents will be asked not to initiate any new psychotherapy for the child during the study
* Subjects may also be excluded after the first MR scan if we are unable to localize the two regions in their brain that are used as targets for the active and control neurofeedback conditions.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms after the intervention compared to baseline | Baseline, 4 days post-NF, 2 weeks post-NF, and 1 month post-NF
  Symptom severity is assessed using the Yale Global Tic Severity Scale (YGTSS) before NF and at several time points in the month following the completion of NF training.

SECONDARY OUTCOMES:
Change in control over activity in the SMA target region during NF compared to baseline | Baseline and during NF
  Control over the SMA is computed as the difference in the blood-oxygenation-level-dependent (BOLD) signal in SMA during up-regulate compared to down-regulate blocks. This measure is computed both in the NF scans and in the control task scans prior to the start of NF. Improvement in control for each subject is the difference of these two (i.e., control during NF minus control during pre-intervention control task scans).

OTHER OUTCOMES:
Changes in resting state functional connectivity to SMA in NF group | Baseline and one month post-NF
  Functional connectivity is measured as temporal synchrony in the BOLD data in functional scans in which participants are just resting in the scanner. These scans are collected at baseline and one month after the neurofeedback training. Connectivity to the SMA will be computed for each time point and the change in the neurofeedback group will be examined and correlated with symptom improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hampson, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the National Institute of Mental Health Data Archive (NDA) and made available to other researchers.
Supporting Information: Study Protocol
Time Frame: Data are uploaded every 6 months to NDA during the trial. Demographic and baseline data are released by NDA four months after upload. Outcome measures are released by NDA upon publication.